CLINICAL TRIAL: NCT02643498
Title: A Dose Escalation Trial of Stereotactic Body Radiotherapy (SBRT) After Induction Chemotherapy for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-109
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
Keywords: Stereotactic Body Radiotherapy (SBRT); 15-109
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): Cohorts 1-3 After completion of induction chemotherapy, stereotactic body radiotherapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
  Cohorts 4-6 For cohort 4, dose prescription will start at 7 Gy x 6 fractions (42Gy, isoeffective to 11 Gy x 3), followed by 4.8 Gy x 12 (54Gy) and 4.5Gy x 15 (67.5Gy).
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT)

SUMMARY:
The purpose of this study is to find out the maximum dose of SBRT that can be safely given after chemotherapy for treatment of pancreatic cancer that cannot be removed surgically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytopathologically confirmed adenocarcinoma of the pancreas.
* Locally advanced, unresectable pancreatic cancer as confirmed by the multidisciplinary input from a hepatobiliary surgeon and as defined on CT as having tumor abutment of >180° (> 50%) of the circumference of the superior mesenteric artery (SMA) or celiac axis, unreconstructable superior mesenteric vein (SMV) or PV involvement.
* No evidence of distant metastasis either prior to or after induction chemotherapy.
* Completion of at least 3 months, but no more than 6 months of standard induction chemotherapy for LAPC, which may include FOLFIRINOX or gemcitabine and nab-paclitaxel, preferably within 2-4 weeks but no longer than 8 weeks.
* Pancreatic tumor size ≤ 5 cm.
* Age ≥18 years
* ECOG 0-1.
* Patients must have acceptable organ and marrow function as defined below:

  * Leukocytes >3,000/uL
  * Absolute neutrophil count >1,500/uL
  * Platelets >50,000/uL
  * Total bilirubin Within 2 x upper limit of normal
  * AST (SGOT)/ALT (SGPT) <2.5 x institutional upper limit of normal
  * Creatinine-Creatinine clearance Within 1.5 x upper limit of normal OR >60 mL/min for patients with creatinine levels above institutional normal
* Ability to understand and follow the breathing instructions involved in the respiratory gating procedure or to tolerate compression sufficient to reduce fiducial motion to ≤ 5mm
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior abdominal radiotherapy.
* Patients receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Contraindication to Magnetic Resonance Imaging
* Patients in which iodine contrast is contraindicated
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 4 weeks after the study are excluded. This applies to any woman who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months, or women on hormone replacement therapy with serum FSH levels greater than 35 mIU/mL. A negative urine or serum pregnancy test must be obtained within 14 days prior to the start of study therapy in all women of child-bearing potential. Male subjects must also agree to use effective contraception for the same period as above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of SBRT | after at least 3 months of induction chemortherapy
  Dose limiting toxicities (DLT) are defined by ≥ Grade 3 treatment-related GI toxicity within 3 months of SBRT. These include: (1) Bowel (includes bowel perforation, obstruction, or hemorrhage) and (2) Stomach (bleeding ulcer, perforation). We will employ a standard 3+3 dose-escalation scheme. Patients will be accrued to the study in cohorts of 3.

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Reyngold, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and follow-up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and follow-up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and follow-up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-up), Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/